CLINICAL TRIAL: NCT04467827
Title: Assessment of Body Posture Connection From the Level and Form of Physical Activity in a Group of Young People
Brief Title: Connection of Body Posture From the Level and Form of Physical Activity in a Group of Young People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Other Study IDs: BW- 2020- SUM
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-05

CONDITIONS: Body Posture
Keywords: body posture, physical activity , young people
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group A1 male: back shape neutral - a vertical line applied to the back of the body meets at the level of the thoracic segment and buttocks
  Interventions: Diagnostic Test: examining group
- Group A2 female: back shape neutral - a vertical line applied to the back of the body meets at the level of the thoracic segment and buttocks
  Interventions: Diagnostic Test: examining group
- Group B1 male: round back shape - a vertical line applied to the back of the body contacts only at the level of the thoracic segment
  Interventions: Diagnostic Test: examining group
- Group B2 female: round back shape - a vertical line applied to the back of the body contacts only at the level of the thoracic segment
  Interventions: Diagnostic Test: examining group
- Group C1 male: round back shape - a vertical line applied to the back of the body only touches the level of the buttock section
  Interventions: Diagnostic Test: examining group
- Group C2 female: round back shape - a vertical line applied to the back of the body only touches the level of the buttock section
  Interventions: Diagnostic Test: examining group

INTERVENTIONS:
Diagnostic Test: examining group — Posture assessment in young healthy people depending on their level of physical activity

SUMMARY:
The assumption of the research is to assess the change in body posture depending on the given level of physical activity in young people. The aim of the study is to assess body posture in young healthy people depending on their level of physical activity. The research will allow the analysis of the correlation between the level of energy expenditure and the occurrence of changes in body posture. The obtained results will allow the development of diagnostic and therapeutic programs for the prevention of overload changes in the spine in young people.

DETAILED DESCRIPTION:
The study will be conducted in a group of 200 people aged 19-25. Posture assessment will concern the measurement of curvatures in the sagittal plane of the spine using a gravitational Rippstein plurimeter and performing a three-dimensional analysis of the spine using the DIERS 3D device. In addition, a modified Matthias test will be performed using the DIERS 3D device, where kyphosis and lordosis parameters in the sagittal plane of the spine at isometric tension of the spinal muscles will be assessed. The spinal motion in the sagittal and frontal planes will also be measured using a digital inclinometer. In the second stage of the study, the participants will participate in the activity in the form of endurance training "Nordic Walking" (NW) for a period of 8 weeks 3 times a week. The recording of energy expenditure during a normal day of activity will be done using an Actigraph GT3X accelerometer. After a period of 8 weeks, all measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* age from 19 to 25 years old
* good health enabling the exercise of various forms of physical effort -cardiologically stable persons, without significant respiratory, nervous and musculoskeletal disorders / no other diseases
* written consent of the examined person

Exclusion Criteria:

* age below 19 and above 25,
* health condition preventing the exercise of various forms of physical effort (cardiologically unstable persons with significant respiratory, nervous and musculoskeletal disorders / other diseases that prevent physical activity,
* lack of written consent of the examined person,
* lack of cooperation of the examined person during the test

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Students of Medical University of Silesia in Katowice, Poland
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-01-27 (Estimated); Study Completion 2023-02-24 (Estimated)

PRIMARY OUTCOMES:
Body posture parameters assessed: | 9 weeks
  * Rippstein plurimeter - measurement of curvature of the spine - kyphosis, lordosis and measurement of the range of spinal mobility in the frontal and transverse planes (ROM)
  * formetric measurement using the DIERS 3D three-dimensional analysis system-tilt of the torso, pelvic lift, pelvic rotation ,pelvic tilt, kyphosis angle, lordosis angle, spine rotation ,side deviation
  * assessment of spinal flexibility (measuring device - digital inclinometer) - range of spinal mobility in the frontal and sagittal plane (ROM)
Physical activity parameters assessed: | 9 weeks
  accelerometer ActiGraph GT3X - assessment of MET energy expenditure and the number of steps performed during one day

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Rehabilitation, Faculty of Health Sciences in Katowice, Medical University of Silesia, Katowice,, Katowice, Katowice Ochojec, Poland

IPD SHARING:
Plan to Share IPD: Undecided